CLINICAL TRIAL: NCT00540410
Title: A Randomized Study to Compare Artesunate + Amiodaquine Versus Artemether + Lumefantrine in the Treatment of Repeated Uncomplicated Plasmodium Falciparum Malaria Attacks Occurring During 2 Years in a Cohort in Senegal
Brief Title: Cohort Study in Senegal Comparing Artesunate + Amiodaquine in the Treatment of Repeated Uncomplicated Plasmodium Falciparum Malaria Attacks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARAMF_L_02873
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Amodiaquine; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Coarsucam® (artésunate (AS) + amodiaquine (AQ) as fixed dose combination)
- 2 (Active Comparator)
  Interventions: Drug: Coartem® (arthemether+ lumefantrine)

INTERVENTIONS:
Drug: Coarsucam® (artésunate (AS) + amodiaquine (AQ) as fixed dose combination) — Infants tablets: AS 25/AQ 67,5 mg Toddlers tablets: AS 50/AQ 135 mg Once daily, dose according to bodyweight range Duration of treatment: 3days Children tablets: AS 100/AQ 270 mg
  Arms: 1
Drug: Coartem® (arthemether+ lumefantrine) — Tablets, 20/120 mg, oral route, twice daily, dose according to bodyweight range.
  Duration of treatment: 3 days
  Arms: 2

SUMMARY:
Primary objective: to demonstrate the non-inferiority of PCR adjusted adequate clinical and parasitological response at D28 of artesunate + amiodaquine versus artemether + lumefantrine, based on the first malaria attack of each subject.

Secondary objectives:

For the first attack: To compare the two groups of treatment in terms of:

* D14 efficacy
* Parasitological and fever clearance
* Clinical and biological tolerability
* Evolution of gametocyte carriage
* Cardiac tolerability (QTc)

For the repeated attacks: To compare the two groups of treatment in terms of:

* D14 and D28 clinical and parasitological effectiveness (PCR adjusted)
* Clinical and biological tolerability
* Proportion of patients without fever at D3
* Proportion of patients without parasite at D3
* Compliance
* Impact on anaemia

During the total follow-up of the cohort: To compare the two groups of treatment in term of:

* Treatment incidence density
* Impact of repeated treatment on clinical and biological safety
* Impact of repeated treatment on hearing capacity

ELIGIBILITY:
Lists of Inclusion and Exclusion criteria:

Inclusion Criteria:

* adults or children weighting more than 5 kg
* axillary temperature >=37.5°C at D0 or history of fever within the previous 24hrs
* confirmed Plasmodium falciparum monoinfection, with parasitemia>1000mcl
* negative urinary pregnancy test for women of child bearing age before each new administration of treatment

Exclusion Criteria:

* presence of any serious or clinical danger sign of malaria: prostration, consciousness disorders, recent and repeated convulsions, respiratory distress, inability to drink, uncontrollable vomiting, macroscopic haemoglobinuria, jaundice, haemorrhagic shock, systolic BP< 70 mmHg in adults or < 50 mmHg in children, spontaneous bleeding, inability to sit or stand
* severe concomitant disease
* allergy to one of the investigational drugs.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2007-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
PCR corrected and uncorrected clinical and parasitological cure rate | at D28 and for the first attack

SECONDARY OUTCOMES:
PCR corrected and uncorrected clinical and parasitological cure rate | at D28 and for the next attacks
Fever and parasitological clearance | first attack
Proportion of afebrile patients and proportion of patients without parasites | at D3 for the following attacks
Clinical tolerability (incidence and intensity of recorded AE) | during the study period
Biological tolerability (Hb, bilirubin, ALAT, Creatinine, Leukocytes, Neutrophils and platelets count) | during the study period
Cardiac tolerability (QTc) for the first attack in patients group aged >= 12 years) | at the time of the first attack
Assessment and evolution of hearing function in patients groupe aged >=12 years | during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Lemeyre, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Dakar, Senegal

REFERENCES:
- [Derived] Ndiaye JL, Faye B, Gueye A, Tine R, Ndiaye D, Tchania C, Ndiaye I, Barry A, Cisse B, Lameyre V, Gaye O. Repeated treatment of recurrent uncomplicated Plasmodium falciparum malaria in Senegal with fixed-dose artesunate plus amodiaquine versus fixed-dose artemether plus lumefantrine: a randomized, open-label trial. Malar J. 2011 Aug 12;10:237. doi: 10.1186/1475-2875-10-237. PMID 21838909